CLINICAL TRIAL: NCT01695538
Title: The Effect of Yoga on Arrhythmia Burden and Quality of Life in Patients With Inappropriate Sinus Tachycardia
Brief Title: Yoga and Rate and Duration of Inappropriate Sinus Tachycardia (IST) Episodes
Acronym: YOGA STAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12946
Record Dates: First submitted 2012-07-05; First posted 2012-09-28 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Inappropriate Sinus Tachycardia
Keywords: Yoga; atrial tachycardia
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga (Experimental): Participants will be asked to practice yoga 3 days per week, at a minimum and encouraged to practice 7 days per week, for 1 year.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — The subjects will be asked to practice Yoga poses at least 3 times a week at home, although daily Yoga will be encouraged. Participants will be trained in breathing exercises, postures and meditation. Each time they practice yoga will be for 1 hour and include breathing exercises, postures and meditation.

SUMMARY:
Inappropriate sinus tachycardia (IST) is an uncommon form of atrial tachycardia. The term "inappropriate" in medicine is commonly defined as a heart rate greater than 100 beats per minute at rest or with minimal physiological challenge. IST is characterized by an increased resting heart rate with an exaggerated response to exercise or stress.

Yoga has been used extensively around the world as an alternative medicine approach in treating numerous chronic and debilitating diseases. Studies have been conducted in various countries to determine the benefits of Yoga as therapy for these chronic diseases. Several studies have confirmed that yoga can reduce anxiety and regulate the stress response.

Studies in the past have shown that Yoga relieves stress, one of the most common triggers for the arrhythmia and increased heart rate in IST. Based on past studies we hypothesize that patients with IST might benefit by practicing yoga. Yoga may also help in better rate and rhythm control with yoga when employed in combination with usual medical arrangement.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with inappropriate sinus tachycardia

Exclusion Criteria:

* Advanced malignancy or severe co-morbidities such as severe heart failure and with life expectancy less than 1 year
* Pregnant women
* Patients with unmedicated or uncontrolled high blood pressure
* Patients with past history of Pnuemothorax
* Patients with severe cervical spondylitis and cervical, thoracic, or lumbar disc prolapse
* Patients with carotid stenosis
* Patients with history of psychosis (evidence of acute episodes with deep and prolonged meditation) or substance abuse
* Patients with history of epilepsy (evidence of acute episodes with deep and prolonged medication)
* Patients with glaucoma
* Patients with history of Total Hip Replacement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Determine if Yoga affects the rate and duration of IST episodes | Change from Baseline to 3 Months
Determine if Yoga affects the rate and duration of IST episodes | Change from Baseline to 1 Year

SECONDARY OUTCOMES:
Effect yoga has on resting heart rate or occurrence of IST episodes in patients that have undergone treatment with medications and/or ablation procedures | 3 Months, 1 Year
Change in Quality of Life | 3 Months, 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, FACC, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States